CLINICAL TRIAL: NCT03363243
Title: Advancing STOP: Self-regulation Therapy for Opioid Addiction and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-1849
Record Dates: First submitted 2017-10-16; First posted 2017-12-06 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Opioid-use Disorder; Chronic Pain
MeSH Terms: conditions — Opioid-Related Disorders; Chronic Pain | interventions — Therapeutics; Population Groups

STUDY DESIGN:
Intervention Model Description: 1 Treatment group with STOP therapy; 1 Treatment as usual group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STOP Therapy Treatment group (Experimental): Self-regulation Treatment for Opioid addiction and Pain (STOP) is a 12-week, rolling entry group therapy protocol that underwent initial development in a previous K23 study. Treatment consists of weekly 90-minute CBT+SR (Self Regulation) treatment with skill building exercises for co-morbid opioid addiction and pain. STOP will be provided in lieu of TAU (Treatment as Usual) group therapy.
  Interventions: Other: STOP Therapy Treatment group
- Treatment as usual (TAU) group (Active Comparator): Psychotherapy for Addiction in conjunction with medication assisted treatment. Standard community treatment for opioid addiction consists of 90-minute weekly rolling entry addiction treatment for 12 weeks to allow for the learning and rehearsal of skills designed to reduce relapse.
  Interventions: Other: Treatment as usual (TAU) group

INTERVENTIONS:
Other: STOP Therapy Treatment group — Testing of the STOP Therapy protocol
  Arms: STOP Therapy Treatment group
Other: Treatment as usual (TAU) group — Treatment as usual in the community through group therapy
  Arms: Treatment as usual (TAU) group

SUMMARY:
The public health relevance of this proposed project is substantial given the current opioid abuse epidemic as identified by the Centers for Disease Control (CDC). This study finalizes and tests a new psychotherapy treatment that is designed to treat chronic pain and opioid addiction at the same time in a format that could be easily used in a community addiction treatment setting. Final products of the study will yield an integrated STOP (Self-regulation/Cognitive-behavioral therapy (CBT) Therapy for Opioid addiction and Pain) manual guided protocol, patient workbook, and therapist training protocol.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years old;
2. Willing to adhere to study protocol including treatment sessions and assessments;
3. Individuals have a history of co-morbid opioid use disorder and chronic pain;
4. Cognitively able to participate and give informed consent.

Exclusion Criteria:

1. Acute or unstable psychotic disorder;
2. Psychiatric hospitalization or suicide attempt in the past 3 months
3. Patient has been diagnosed with an unstable cardiovascular condition including: myocardial infarction, arrhythmia, or poorly controlled hypertension in the past 3 months
4. Lack of verbal and written English fluency
5. Over the age of 65 since evidence suggests pain perception alters with age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-04-21 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in Daily Functioning - Pain | Baseline (week 1) to post-treatment assessment time-point (week 14) and to a 1-month post-treatment follow-up assessment for each participant (approximately 4-5 month total time frame per participant)
  Multi-dimensional pain inventory - 60 items (participant ratings 0 to 6 on various measures, from none to extreme or from never to very often, related to their pain and functioning); subscales (ratings in each subscale are averaged to form subscale scores): Interference, Support, Pain Severity, Life-Control, Affective Distress, Negative Responses, Solicitous Responses, Distracting Responses, Household Chores, Outdoor Work, Activities Away from Home, Social Activities, General Activity

SECONDARY OUTCOMES:
Changes in Substance Use | Baseline (week 1), then assessed weekly over the course of the therapy treatment (approximately 4-5 months for each participant)
  urinalysis toxicity screening

OTHER OUTCOMES:
Substance Use, self-report | Weekly through study completion, approximately 4-5 months for each participant
  Timeline Follow back self report (Report alcohol/drug that you may have used in the past two weeks)
Pain assessment through Cold Pressor task | Assessed at initial session (week 1), follow up (~12-13 weeks after initial session) and 1 month follow up (~4-5 months after initial session) for each participant
  Cold pressor task assessment measures: 0-100 acute pain levels after task (0 being no pain, 100 being extreme pain), pain sensitivity (duration in water until reported feeling pain), pain tolerance (length of time hand is kept in cold water), physiological response to cold water
Daily Functioning - Timed up and go | Assessed at initial session (week 1), follow up (~12-13 weeks after initial session) and 1 month follow up (~4-5 months after initial session) for each participant
  Timed up and go test - measure of function with correlates to balance and fall risk; participant is timed while getting up from a chair, walking, and returning to a seated position; scores of greater than or equal to 14 seconds indicate higher fall risk.
Daily functioning - physical performance | Assessed at initial session (week 1), follow up (~12-13 weeks after initial session) and 1 month follow up (~4-5 months after initial session) for each participant
  Modified Physical performance test - 9 items in which participant performs basic physical activities: Standing Static Balance, Chair rise, Lift book, Put on jacket, Pick up penny, turn 360 degrees, 50 ft walk test, climb one flight of stairs, climb stairs (max. 4 flights); items are scored 0 to 4 based on time to complete task (with 0 being unable to complete task, 1 being longest timeframe to complete task and 4 being shortest timeframe)
Current pain levels | Weekly through study completion, approximately 4-5 months for each participant
  0-100 Current pain rating scale (with 0 being no pain, 100 being extreme pain)
Self-efficacy - Drug abstinence | Assessed at initial session (week 1), follow up (~12-13 weeks after initial session) and 1 month follow up (~4-5 months after initial session) for each participant
  Drug abstinence self-efficacy scale - 12 items, 1-5 scale (1 being not at all confident, 5 being extremely confident)
Pain Catastrophizing | Assessed at initial session (week 1), follow up (~12-13 weeks after initial session) and 1 month follow up (~4-5 months after initial session) for each participant
  Pain Catastrophizing scale - assesses 13 items on a 0-4 scale (0-not at all, 1-to a slight degree, 2-to a moderate degree, 3-to a great degree, or 4-all the time)
Self-efficacy - Pain | Assessed at initial session (week 1), follow up (~12-13 weeks after initial session) and 1 month follow up (~4-5 months after initial session) for each participant
  Pain self-efficacy questionnaire - 10 items, 0-6 scale (0 - not at all confident, 6 - extremely confident)
Craving - Brief Substance Craving Inventory | assessed at initial session (week 1), follow up (~12-13 weeks after initial session) and 1 month follow up (~4-5 months after initial session) for each participant
  Brief Substance Craving Inventory - self-report of drug cravings within the past 24 hours
Craving - Current Craving levels | assessed weekly from 2nd week through 13th week for each participant
  Desire for Drug and current craving levels questionnaire - 14 items, 1-7 scale (1-not at all, 7- very much)
Distress Tolerance Scale | assessed at initial session (week 1), follow up (~12-13 weeks after initial session) and 1 month follow up (~4-5 months after initial session)
  Distress tolerance scale - 15 items, rate from "strong agree" to "strong disagree"
Coping | assessed at initial session (week 1), follow up (~12-13 weeks after initial session) and 1 month follow up (~4-5 months after initial session) for each participant
  Brief Cope Inventory - items rated from "never" to "always" on 28 items related to coping
Positive and Negative Affect Scale | assessed weekly from 2nd week through 13th week for each participant
  PANAS - ratings for how a participant has felt in the past two weeks, from 1 ("very slightly or not at all") to 5 ("extremely")
Addiction Severity Index | assessed at initial session (week 1)
  ASI - survey on participant's baseline addiction severity; 5 parts (Background, Basic Health, Relationships, Alcohol and Drug Use, Legal situation)
Hospital Anxiety and Depression scale | assessed at initial session (week 1), follow up (~12-13 weeks after initial session) and 1 month follow up (~4-5 months after initial session) for each participant
  HADS - asks participants to indicate how they generally feel on 14 items
Session feedback | weekly through study completion, approximately 4-5 months for each participant
  12 items, 1 for each weekly therapy topic, participants rate from 1 (very useful and will definitely use the strategies discussed) to 4 (not very useful and may not use the strategies discussed)
Weekly attendance data sheet | weekly through study completion, approximately 4-5 months for each participant
  table indicating which participants and the total number of participants that attend the therapy group each week
Eligibility phone screening | assessed at initial session (week 1) for each participant
  6 yes or no items for inclusion/exclusion criteria, 1 open-ended item to provide medication and dosage frequency, 1 item to provide typical pain level on 0-10 scale
Demographics data sheet | assessed at initial session (week 1) for each participant
  demographics information

CONTACTS AND LOCATIONS:
Overall Officials: Amy B Wachholtz, PhD, MDiv, MS, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wachholtz A, Robinson D, Epstein E. Developing a novel treatment for patients with chronic pain and Opioid User Disorder. Subst Abuse Treat Prev Policy. 2022 May 7;17(1):35. doi: 10.1186/s13011-022-00464-4. PMID 35525964